CLINICAL TRIAL: NCT04641624
Title: Soluble Fms-like Tyrosine Kinase-1, Proangiogenic Protein Placental Growth Factor, and Niacin Levels in Women With Premature Ovarian Insufficiency
Brief Title: sFlt- 1, PIGF, and Niacin Levels in Women With Premature Ovarian Insufficiency
Acronym: POİ&niacin
Status: Completed | Type: Observational
Sponsor: Cengiz Gokcek Women's and Children's Hospital (Other)
Responsible Party: Principal Investigator, Ali Ovayolu, Principal Investigator, Cengiz Gokcek Women's and Children's Hospital
Other Study IDs: CengizGWCH11
Record Dates: First submitted 2020-11-18; First posted 2020-11-24 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Premature Ovarian Insufficiency
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Premature ovarian insufficiency (POI): POI is a clinical syndrome defined by loss of ovarian activity before the age of 40 years. POI is characterized by menstrual disturbance (amenorrhea or oligomenorrhea) with raised gonadotrophins and low estradiol.
  The study population will be consisted of 45 women with POI as study group.
  Interventions: Other: ultrasound assessment
- Control group: 45 patients with normal healthy women as control group.
  Interventions: Other: ultrasound assessment

INTERVENTIONS:
Other: ultrasound assessment — soluble fms-like tyrosine kinase-1, proangiogenic protein placental growth factor, and niacin measurementswith a commercially available enzyme-linked immunosorbent assay (ELISA) kit.
  Other Names: soluble fms-like tyrosine kinase-1, proangiogenic protein placental growth factor, and niacin measurements

SUMMARY:
Aim: To evaluate serum soluble fms-like tyrosine kinase-1, proangiogenic protein placental growth factor, and niacin levels in women with premature ovarian insufficiency (POI) and to compare the results with those of healthy subjects.

Methods: This prospective study will be included 45 women with idiopathic premature ovarian insufficiency and 45 controls. The blood for analysis will be obtained at the early follicular phase of the menstrual cycle and serum soluble fms-like tyrosine kinase-1, proangiogenic protein placental growth factor, and niacin levels will be measured using a commercially available ELISA kit.

DETAILED DESCRIPTION:
This will be an observational prospective cohort study conducted at Obstetrics and Gynecology Department of Cengiz Gokcek Obstetrics and Children's Hospital between November 2020 and April 2021. The investigators will be recruited 45 subjects with idiopathic POI, and 45 healthy patients were selected for the control group. All patients will be given their oral and written informed consent before their inclusion in the study. The protocol was approved by the Ethics Committee for Clinical Research of Gaziantep University (Reference number: 2020/320). The study strictly will be adhered to the principles of the Declaration of Helsinki.

Women between the ages of 18-39 will be included. A volunteer group of healthy women who will be visited the gynecology clinic for routine examinations and women who will be admitted for pre-pregnancy tests will be invited randomly to this research as a control group. Healthy women, who will be returned during their early follicular phase of the menstrual cycle, will be recruited as the control group subjects. The exclusion criteria will be as follows: women with evidence for karyotypic, metabolic, toxic, or iatrogenic cause of the ovarian insufficiency and any women who use any medication for POI treatment. At enrollment, for both groups, the investigators will be collected data about age, height, weight, BMI, age of menarche, obstetrics history, history of smoking, regular exercise and family history of POI. At enrolment, all patients will be underwent vaginal ultrasonography for the assessment of antral follicle count (AFC) and venous blood sample from the antecubital veins for measuring serum concentration of soluble fms-like tyrosine kinase-1, proangiogenic protein placental growth factor, and niacin, Follicle-stimulating hormone (FSH), E2, anti-mullerian hormone (AMH) and complete blood count (CBC). In control subjects venous blood samples and AFC will be collected during the early follicular phase of the menstrual cycle. The serum samples will be stored in aliquots at -80°C prior to the analyses of sFlt- 1, PIGF, and niacin. The serum soluble fms-like tyrosine kinase-1, proangiogenic protein placental growth factor, and niacin level will be measured using a commercially available enzyme-linked immunosorbent assay (ELISA) kit. Then, this study will be determined maternal serum soluble fms-like tyrosine kinase-1, proangiogenic protein placental growth factor, and niacin levels in women with POI (n=45) compared to those of volunteer healthy women (n=45). Then, these three markers levels will be compared in both group.

ELIGIBILITY:
Inclusion Criteria:

* women with POI
* Healthy women

Exclusion Criteria:

1. women with any systemic condition (such as chronic hypertension, renal disease)
2. history of using any medication
3. drug user
4. history/presence of malignancy
5. history of Radiotherapy/chemotherapy
6. polycystic ovary syndrome
7. women who had any other acute/chronic infection or fever
8. Patients whose chromosome analysis result is not normal
9. history of ovarian surgery
10. Ovarian cysts/mass
11. pregnancy
12. lactation

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — POI is a clinical syndrome defined by loss of ovarian activity before the age of 40 years. POI is characterized by menstrual disturbance (amenorrhea or oligomenorrhea) with raised gonadotrophins and low estradiol. It is estimated to affect 1% of women under the age of 40, 0.1% under 30 and 0.01% under 20.
Study Population: The investigators consecutively will be recruited 45 subjects with POI, and 45 healthy women will be selected for the control group.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
sFlt- 1 levels | 1 week
  The primary outcome measure in this analysis will compare sFlt- 1 levels in the idiopathic POI group and control group.
PIGF levels | 1 week
  The primary outcome measure in this analysis will compare PIGF levels in the idiopathic POI group and control group.
niacin levels | 1 week
  The primary outcome measure in this analysis will compare niacin levels in the idiopathic POI group and control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Cengiz Gokcek Women's and Child's hospital, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] European Society for Human Reproduction and Embryology (ESHRE) Guideline Group on POI; Webber L, Davies M, Anderson R, Bartlett J, Braat D, Cartwright B, Cifkova R, de Muinck Keizer-Schrama S, Hogervorst E, Janse F, Liao L, Vlaisavljevic V, Zillikens C, Vermeulen N. ESHRE Guideline: management of women with premature ovarian insufficiency. Hum Reprod. 2016 May;31(5):926-37. doi: 10.1093/humrep/dew027. Epub 2016 Mar 22. PMID 27008889
- [Result] Wang S, Sun M, Yu L, Wang Y, Yao Y, Wang D. Niacin Inhibits Apoptosis and Rescues Premature Ovarian Failure. Cell Physiol Biochem. 2018;50(6):2060-2070. doi: 10.1159/000495051. Epub 2018 Nov 9. PMID 30415247
- [Result] Maclaran K, Horner E, Panay N. Premature ovarian failure: long-term sequelae. Menopause Int. 2010 Mar;16(1):38-41. doi: 10.1258/mi.2010.010014. No abstract available. PMID 20424285
- [Result] Taraseviciene V, Grybauskiene R, Maciuleviciene R. sFlt-1, PlGF, sFlt-1/PlGF ratio and uterine artery Doppler for preeclampsia diagnostics. Medicina (Kaunas). 2016;52(6):349-353. doi: 10.1016/j.medici.2016.11.008. Epub 2016 Nov 29. PMID 27940029
- [Derived] Ovayolu A, Bostancieri N. A prospective and comparative investigation of blood sFlt-1, P1GF, and niacin concentrations in women with premature ovarian insufficiency. J Obstet Gynaecol Res. 2023 Apr;49(4):1198-1205. doi: 10.1111/jog.15554. Epub 2023 Jan 22. PMID 36682889

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/24/NCT04641624/Prot_SAP_000.pdf